CLINICAL TRIAL: NCT03368040
Title: Comparison Between Tcore(TM) Temperature Monitoring System and Invasive Blood Temperature Measurements
Brief Title: Comparison Between Non-invasive Heat-flux and Invasive Core Temperature Monitoring
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Martin Soehle, Vice head of Anesthesiology, University Hospital, Bonn
Other Study IDs: TCO
Record Dates: First submitted 2017-01-24; First posted 2017-12-11 (Actual); Last update posted 2019-03-29 (Actual); Status verified 2019-03

CONDITIONS: Body Temperature Changes
Keywords: body core temperature
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Tcore — Monitoring system to measure body temperature based on heat-flux technology

SUMMARY:
The body core temperature drops during general anesthesia. To maintain homeostasis, patients require warming measures. Different methods to measure body core temperature exist, which are either highly accurate but invasive, or non-invasive but non-accurate. A new monitoring device, Tcore(TM), enables a non-invasive but accurate core temperature assessment.

This study is performed to quantify accuracy and bias of the Tcore system in comparison with the blood temperature, which is the gold standard of core temperature measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive femoral artery temperature monitoring

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that undergo major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Bias of heat-flux temperature monitoring [%] | from insertion of thermometers to end of surgery
  Over the time course of surgery, the body core temperature is actually measured in the bloodstream (Tbl) and estimated by the heat-flux thermometer (Thf). The bias or median prediction error (MPE) is calculated as median of PE, which is (Tbl-Thf)/Tbl.

SECONDARY OUTCOMES:
Inaccuracy of heat-flux temperature monitoring [%] | from insertion of thermometers to end of surgery
  Over the time course of surgery, the body core temperature is actually measured in the bloodstream (Tbl) and estimated by the heat-flux thermometer (Thf). The inaccuracy or median absolute prediction error (MAPE) is calculated as median of abs(PE), which is (Tbl-Thf)/Tbl.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Bonn, Germany

IPD SHARING:
Plan to Share IPD: No